CLINICAL TRIAL: NCT07272291
Title: A Prospective, Single-Arm Phase II Study of Toripalimab Plus Chemotherapy and Low-Dose Radiotherapy as Neoadjuvant Treatment for Neoadjuvant Therapy-Refractory Esophageal Squamous Cell Carcinoma
Brief Title: A Phase II Study of Toripalimab Plus Chemotherapy and Low-Dose Radiotherapy for Neoadjuvant Therapy-Refractory Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-TCR-2025
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — After 2 cycles of neoadjuvant therapy with stable disease (SD) in efficacy assessment, subjects will sign the informed consent form. Baseline assessment is conducted within 4 weeks before enrollment.
  Enrolled patients first receive low-dose radiotherapy (1.2 Gy × 5), then continue with 2 cycles of the chemotherapy regimen combined with toripalimab (240 mg, once every 3 weeks), followed by surgical treatment.
  Subsequently, based on pathological results:
  Non-pCR patients receive toripalimab monotherapy until disease recurrence, intolerable toxicity, or subject's withdrawal of informed consent. The total duration of study drug administration is at most 1 year, whichever comes first.
  pCR patients directly undergo regular post-surgical survival follow-up.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of neoadjuvant toripalimab combined with chemotherapy and low-dose radiotherapy in patients with esophageal squamous cell carcinoma who are insensitive to neoadjuvant therapy. The main question it aims to answer is:

• Whether adding low dose radiotherapy can improve the efficacy of immunotherapy combined chemotherapy in neoadjuvant setting?

Participants will receive low-dose radiotherapy (1.2 Gy/fraction, 5 fractions), followed by 2 cycles of chemotherapy plus toripalimab (240 mg, q3w). 6 to 8 weeks after treatment completion, a systematic preoperative assessment is conducted, then surgery is performed. Postoperatively, management depends on pathological results:

Non-pathological complete response (non-pCR) patients: Toripalimab monotherapy continues until disease recurrence, intolerable toxicity, informed consent withdrawal, or for 1 year (whichever comes first).

Pathological complete response (pCR) patients: Directly undergo regular postoperative survival follow-up

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 18 years;
* Esophageal cancer staged as T1-4aN1-3M0 or T3-4aN0M0 (per AJCC 8th edition), with histologically confirmed predominant squamous cell carcinoma at initial diagnosis;
* Subjects must complete 2 cycles of preoperative neoadjuvant immunotherapy combined with chemotherapy (any regimen) before enrollment, followed by imaging assessment showing stable disease (SD);
* ECOG performance status score of 0 or 1;
* All required baseline laboratory tests must be completed, with results obtained within 14 days before enrollment. Laboratory tests resluts must meet the following criteria (per CTCAE v5):

WBC ≥ 2000/μL Neutrophils ≥ 1500/μL Platelets ≥ 100 × 10³/μL Hemoglobin ≥ 9.0 g/dL Creatinine: Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance > 50 mL/min (per Cockcroft/Gault formula) AST ≤ 3 × ULN, ALT ≤ 3 × ULN Total bilirubin ≤ 1.5 × ULN (except subjects with Gilbert syndrome, for whom total bilirubin must be < 3 × ULN);

* Tumor tissue and blood must be provided for biomarker analysis. If the provided tumor tissue is insufficient for analysis, additional archived tumor tissue (blocks and/or sections) must be obtained;
* Subjects voluntarily participate in the study, sign a written informed consent form, and are compliant with follow-up;
* Subjects must be willing and able to adhere to scheduled visits, treatment plans, laboratory tests, tumor biopsies, and other study requirements;
* Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days before enrollment, and agree to use effective contraception during the study and for at least 6 months after the last dose of toripalimab. Males with partners of childbearing potential must agree to use effective contraception during the study and for at least 6 months after the last dose.

Exclusion Criteria:

* Subjects with a history of other malignant tumors are excluded, unless complete remission was achieved at least 5 years prior to study entry and no additional treatment is required or anticipated during the study period. Exceptions include, but are not limited to, basal or squamous cell carcinoma of the skin, superficial bladder cancer, or in situ carcinoma of the prostate, cervix, or breast.
* Subjects with known or suspected active autoimmune diseases are excluded. However, enrollment is permitted for subjects with type 1 diabetes, hypothyroidism requiring only hormone replacement therapy, cutaneous conditions not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia), or conditions not expected to recur in the absence of external triggers.
* Subjects who required systemic treatment with corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive agents within 14 days prior to study drug administration are excluded. Inhaled or topical steroids, as well as adrenal replacement steroids, at doses exceeding 10 mg daily prednisone equivalent are allowed only in the absence of active autoimmune disease.
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity are excluded.
* All toxicities attributable to prior anticancer therapy (except nephropathy, neuropathy, hearing loss, alopecia, and fatigue) must resolve to Grade 1 (per NCI CTCAE Version 5) or baseline before study drug administration. Subjects with toxicities from prior anticancer therapy that are not expected to resolve and result in permanent sequelae (e.g., peripheral neuropathy following platinum-based therapy) are permitted, provided the peripheral neuropathy resolves to Grade 2 (per NCI CTCAE Version 5).
* Subjects with any severe or uncontrolled medical condition or active infection that, in the investigator's judgment, may increase the risks of study participation or study drug administration, or impair the subject's ability to complete treatment per the protocol are excluded.
* Subjects with a known positive human immunodeficiency virus (HIV) test result or a confirmed diagnosis of acquired immunodeficiency syndrome (AIDS) are excluded.
* Subjects who received live/attenuated vaccines within 30 days prior to the first study treatment are excluded.
* Subjects with active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection are excluded, including those with: acute or chronic active hepatitis B/ C; HBV DNA >2000 IU/mL or 10⁴ copies/mL; HCV RNA >10³ copies/mL; or concurrent positivity for hepatitis B surface antigen (HBsAg) and anti-HCV antibodies.
* Subjects with a history of allergy or hypersensitivity to any component of the study drug, or a history of severe hypersensitivity to any monoclonal antibody are excluded.
* Subjects currently participating in other interventional clinical studies are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) rate | up to 12 months
  MPR rate is defined as the proportion of participants who have achieved major pathological response（on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy and underwent surgery.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 5 years
  defined as the period from the start of the study treatment to loss of follow-up or death
Pathological Complete Response (pCR) rate | up to 12 months
  Defined as the proportion of patients in postoperative pathology who have no residual live tumor cells in the primary tumor bed or in all excised lymph nodes.
Event Free Survival (EFS) | up to 5 years
  EFS is defined as the time from the start of the study treatment to any of the following events (whichever occurs first): the investigator assessed the disease progression based on imaging according to RECIST 1.1 and therefore was unable to receive curative surgery, local or distant recurrence, or death from any cause.

IPD SHARING:
Plan to Share IPD: No